CLINICAL TRIAL: NCT02805244
Title: A Phase 1, Open-label, Single Dose, Mass Balance Study to Evaluate the Pharmacokinetics, Biotransformation and Excretion of 14C-JTZ-951 in Male Subjects With End-stage Renal Disease Receiving Hemodialysis
Brief Title: Mass Balance Study of JTZ-951 in Subjects With End-stage Renal Disease on Hemodialysis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Akros Pharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: AZ951-U-15-010
Record Dates: First submitted 2016-06-15; First posted 2016-06-17 (Estimated); Last update posted 2016-11-29 (Estimated); Status verified 2016-11

CONDITIONS: Anemia of Chronic Kidney Disease
Keywords: JTZ-951; Pharmacokinetics; 14C-JTZ-951; Mass balance; Time course
MeSH Terms: interventions — enarodustat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- JTZ-951, 14C-JTZ-951 (Experimental): Single oral administration on Day 1; 10 mg JTZ-951, 100 μCi of 14C-JTZ-951
  Interventions: Drug: JTZ-951, 14C-JTZ-951

INTERVENTIONS:
Drug: JTZ-951, 14C-JTZ-951

SUMMARY:
A mass balance study to determine the routes and rates of elimination of radioactivity, to determine total radioactivity in plasma and whole blood over time and compare levels to JTZ-951 and drug-derived entities in plasma and to determine pharmacokinetic (PK) parameters of JTZ-951 and its metabolite(s).

ELIGIBILITY:
Inclusion Criteria:

* Subjects with end stage renal disease on hemodialysis
* Post-dialysis body weight >45.0 kg
* BMI between 18.0 and 40.0 kg/m2 (inclusive)

Exclusion Criteria:

* Subjects with aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >2.0 × upper limit of normal (ULN), or total bilirubin >1.5 × ULN at the Screening Visit
* Subjects who have hepatobiliary disease or condition (such as biliary cirrhosis)
* Subjects with positive test results for HBsAg (hepatitis B surface antigen), HCV antibody or HIV antibody
* Subjects with known history of liver failure or liver surgery
* Subjects with a history or current clinically significant chronic or acute blood loss

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2016-06; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Radioactivity concentration in urine, feces and dialysate | maximum 20 days
Radioactivity concentration in whole blood and plasma | maximum 20 days
Plasma concentrations of JTZ-951 and its metabolite | maximum 20 days
Cmax (maximum concentration) | maximum 20 days
tmax (time to reach maximum concentration) | maximum 20 days
AUC (area under the concentration-time curve) | maximum 20 days
t1/2 (elimination half-life) | maximum 20 days
Number of adverse events | maximum 20 days

CONTACTS AND LOCATIONS:
Locations (1):
- Minneapolis, Minnesota, United States